CLINICAL TRIAL: NCT02292914
Title: Prospective Analysis of Robot-Assisted Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto do Cancer do Estado de São Paulo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NP433/13
Record Dates: First submitted 2014-09-03; First posted 2014-11-18 (Estimated); Last update posted 2019-08-08 (Actual); Status verified 2019-08

CONDITIONS: Esophageal Cancer; Gastric Cancer; Pancreatic Cancer; Rectal Cancer; Bladder Cancer; Prostate Cancer; Renal Cancer; Uterus Cancer; Head and Neck Cancer; Lung Cancer
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms; Pancreatic Neoplasms; Rectal Neoplasms; Urinary Bladder Neoplasms; Prostatic Neoplasms; Kidney Neoplasms; Uterine Neoplasms; Head and Neck Neoplasms; Lung Neoplasms | interventions — Robotic Surgical Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Robot-Assisted Surgery (Experimental): patients undergoing robot assisted surgery for the treatment of cancer
  Interventions: Procedure: Robot-assisted surgery
- Conventional Surgery (Active Comparator): patients undergoing conventional surgery for the treatment of cancer
  Interventions: Procedure: Conventional Surgery

INTERVENTIONS:
Procedure: Robot-assisted surgery — Robot-assisted esophagectomy; Robot-assisted subtotal gastrectomy; Robot-assisted pancreatectomy;Robot-assisted rectal resection; Robot-assisted radical cistectomy;Robot-assisted prostatectomy;Robot-assisted Partial Nephrectomy; Robot-assisted hysterectomy;Robot-assisted Resection of malignant tumors of the mouth and orofaringolaringe; Robot-assisted lung lobectomy
  Arms: Robot-Assisted Surgery
Procedure: Conventional Surgery — Thoracoscopic Esophagectomy; Open rectal resection and rectal laparoscopy resection; Open radical cistectomy; Open prostatectomy; Open Partial Nephrectomy; Laparoscopic hysterectomy; Laparoscopic lung lobectomy
  Arms: Conventional Surgery

SUMMARY:
The robot-assisted surgery allows three-dimensional view, detailed access of small structures, depth perception and articulated movements with wide latitude. Thinking about the inclusion of this branch of surgical outcome ICESP encouraged the training of their doctors and other health professionals , and has three tutors in the area of robot- assisted laparoscopic surgery , and various medical clinical staff , already trained , and already perform the procedure in other centers . The da Vinci ® Surgical System ( only existing in the World market) , consisting of one or two consoles for the surgeon and a tutor if necessary was adopted. Ergonomically designed, a stand next to the patient , with four interactive robotic arms , one of them , a vision system for high performance and the other three for exclusive EndoWrist ® instruments . Driven by the latest robotic technology , computer programs , frictionless transmission of manual controls , movements in scale and filtered made by the surgeon in the da Vinci ® System console are translated into precise movements of the instruments EndoWrist ® For surgeons , the da Vinci ® System offers superior 3D viewing with larger surgical precision ergonomic comfort and dexterity . For hospitals , the da Vinci ® Surgical System enables clinical and economic benefits of minimally invasive surgery are applied to a broader base of patients cirúrgicos.The main objective is to evaluate the safety and effectiveness of robotic surgery in the surgical treatment of cancer in operations below, as their specialties : Digestive , Urology , Gynecology , Head and Neck and Thorax . This is a prospective study lasting 36 months , where 1120 patients with surgical diseases in programming for the following operations will be studied : transthoracic esophagectomy ; subtotal gastrectomy with lymphadenectomy ; partial pancreatectomy ; resection of the rectum ; prostatectomy ; cystectomy ; partial nephrectomy ; hysterectomy with or without pelvic and paraaortic lymphadenectomy ; resection of malignant tumors of the mouth and orofaringolaringe and lung lobectomy . Patients will come from the outpatient services of the Institute of Cancer of São Paulo - ICESP

DETAILED DESCRIPTION:
This is a prospective study lasting 36 months. This project includes 10 subprojects in five different specialties:

Specialty: Surgery of the Digestive System Subproject 1: trans-thoracic esophagectomy Subproject 2: subtotal gastrectomy with lymphadenectomy Subproject 3: partial pancreatectomy Subproject 4: resection of the rectum Specialty: Urology Surgery Subproject 5: cystectomy Subproject 6: Prostatectomy Subproject 7: Partial Nephrectomy Specialty: Gynecological Surgery Activity 8: Hysterectomy with or without pelvic lymphadenectomy and paraaortic Specialty: Head and Neck Surgery Activity 9: resection of malignant tumors of the mouth and orofaringolaringe Specialty: Thoracic Surgery Subproject 10: pulmonary lobectomies

Each subproject will have a study design, inclusion criteria, exclusion criteria and specific methodologies.

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible for robotic-assisted surgery

Exclusion Criteria:

* Pregnant patients
* Patients with decompensated systemic diseases
* Patients who were unfit for general anesthesia
* Patients without an indication for surgical treatment of cancer

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1120 (Estimated)
Dates: Start 2014-03-10; Primary Completion 2020-07-10 (Estimated); Study Completion 2020-07-10 (Estimated)

PRIMARY OUTCOMES:
Postoperative Complications | 30 days
  The postoperative complications will be mesured by clavien-dindo scale

SECONDARY OUTCOMES:
ICU and hospital length of stay | 2 days

OTHER OUTCOMES:
Surgical time | 1 day
Intraoperative complications | 1 day
  The intraoperative complications will be mesured by clavien-dindo scale
quality of life of cancer patients | 36 months
  The quality of life will be measured by the EORTC QLQ-C30 questionnaire, developed to assess the quality of life of cancer patients
overall survival | 5 years
Disease free survival | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Cecconello, MD, Principal Investigator — Faculdade de Medicina da USP; Ulysses Ribeiro-Junior, MD, Principal Investigator — Faculdade de Medicina da USP
Locations (1):
- Instituto do Câncer de São Paulo - ICESP, São Paulo, Brazil

REFERENCES:
- [Derived] Abdalla RZ, Nahas WC, Cecconello I, Ribeiro U Jr. Prospective study of a structured robotic surgery training program in a public cancer hospital in Brazil. J Robot Surg. 2025 Oct 16;19(1):695. doi: 10.1007/s11701-025-02881-6. PMID 41099765
- [Derived] Nahas WC, Rodrigues GJ, Rodrigues Goncalves FA, Sawczyn GV, Barros GG, Cardili L, Guglielmetti GB, Fazoli AJC, Cordeiro MD, Cassao VDA, Chade DC, Neves De Oliveira LC, Murta CB, Pontes Junior J, Trindade EM, Bastos DA, Sarkis AS, Mitre AI, Trinh QD, Coelho RF. Perioperative, Oncological, and Functional Outcomes Between Robot-Assisted Laparoscopic Prostatectomy and Open Radical Retropubic Prostatectomy: A Randomized Clinical Trial. J Urol. 2024 Jul;212(1):32-40. doi: 10.1097/JU.0000000000003967. Epub 2024 May 9. PMID 38723593
- [Derived] Ribeiro U Jr, Dias AR, Ramos MFKP, Yagi OK, Oliveira RJ, Pereira MA, Abdalla RZ, Zilberstein B, Nahas SC, Cecconello I. Short-Term Surgical Outcomes of Robotic Gastrectomy Compared to Open Gastrectomy for Patients with Gastric Cancer: a Randomized Trial. J Gastrointest Surg. 2022 Dec;26(12):2477-2485. doi: 10.1007/s11605-022-05448-0. Epub 2022 Sep 20. PMID 36127557
- [Derived] Terra RM, Araujo PHXN, Lauricella LL, Campos JRM, Trindade JRM, Pego-Fernandes PM. A Brazilian randomized study: Robotic-Assisted vs. Video-assisted lung lobectomy Outcomes (BRAVO trial). J Bras Pneumol. 2022 Jul 8;48(4):e20210464. doi: 10.36416/1806-3756/e20210464. eCollection 2022. PMID 35830078